CLINICAL TRIAL: NCT06021899
Title: Effects of Classic Constraint Induced Movement Therapy and Its Modified Form on Quality of Life of Children With Hemiplegic Cerebral Palsy
Brief Title: Effects of Classic and Modified CIMT on Quality of Life of Children With Hemiplegic CP
Acronym: CIMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Education Research Foundation (HERF) (Other)
Responsible Party: Principal Investigator, Mamoona Tasleem Afzal, Mamoona Tasleem Afzal, Health Education Research Foundation (HERF)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YIRS/007
Record Dates: First submitted 2023-08-26; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: Constraint induced movement therapy; Cerebral palsy; CPQOL
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classic CIMT group (Active Comparator): Total session of 6 hours a day, 5 days per week for 3 weeks to Classic CIMT groups will be given.
  Interventions: Other: modified constraint induced movement therapy
- mCIMT group (Experimental): Session of 6 hours a day, 5 session per week for first 2 weeks (CIMT), session of 2 hours a day, 5 days per week for last 1 week (BIT) to modified CIMT group will be given.
  Interventions: Other: modified constraint induced movement therapy

INTERVENTIONS:
Other: modified constraint induced movement therapy — Modified CIMT protocol that was based on suggestions made by Dromerick, Edwards, and Hahn (2000) . Modifications were reductions in the duration of mitt wear and massed practice compared with the traditional protocol
  Other Names: classic constaint induced movement therapy

SUMMARY:
The purpose of this research is to see the effect of classic constraint-induced movement therapy and its modified form on quality of life of children with hemiplegic cerebral palsy. Randomized controlled trials with 2-3 weeks follow-up. The sample size is 40. The subjects are divided in two groups, 20 subjects in classical CIMT group and 20 in modified CIMT group. Study duration is of 6 months. Sampling technique applied will be purposive non probability sampling technique. Only 4-12 years individual with hemiplegic cerebral palsy are included. Tools used in the study are Cerebral palsy (quality of life) and Kid Screen 27.

DETAILED DESCRIPTION:
Both CCIMT and MCIMT are effective treatments to improve quality of life of children with CP. However conflicting evidence is present on which one of these is more effective and no final conclusion can be made to date. This study intends to add to the literature and contribute in reaching final conclusion about the superiority of either intervention. The purpose of this study was to see the psychosocial effect (quality of life) of CIMT and its modified form on HCP

ELIGIBILITY:
Inclusion Criteria:

* 4 to 12 years CP with unilateral, bilateral or severely asymmetrical impairment Manual Ability Classification System(MACS) I, II or III Wrist extension capacity at least 20°; fingers with 10° of complete flexion Children able to follow Command

Exclusion Criteria:

* Children also having disabilities other than Cerebral palsy Contractures that significantly limit functional arm use. Children with MR

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Cerebral Palsy Quality of Life CP(QOL) | 3 weeks.
  The Cerebral Palsy Quality of Life for Children (CP QOL-Child) is the first health condition-specific questionnaire designed for measuring QOL in children with cerebral palsy (CP) aged 4-12 years. CP QOL Questionnaires measure include : Social wellbeing & acceptance, Feelings about functioning, Participation & physical health, Emotional wellbeing & self-esteem, Access to services, Pain & impact of disability, Family health

SECONDARY OUTCOMES:
Kid Screen 27 | 3 weeks
  The KIDSCREEN-27 was developed as a shorter version of the KIDSCREEN-52 with a minimum of information loss and with good psychometric properties. The KIDSCREEN-27 with five dimensions resulted. All five dimensions are Rasch scales: Physical Well-Being (5 items), Psychological Well-Being (7 items), Autonomy & Parents (7 items), Peers & Social Support (4 items), and School Environment (4 items)

CONTACTS AND LOCATIONS:
Overall Officials: Saad Tariq, master, Principal Investigator — Riphah International University
Locations (1):
- Yusra Institute of Rehablitation Science, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No